Enhancing Skin Cancer Early Detection and Treatment in Primary Care

NCT05675709

## March 1, 2025

Final approach to analysis

## **Analyses**

We used descriptive analyses to examine participating clinician characteristics and rates of e-consults, dermatology referrals and biopsies performed (defined as the number of cases per 1000 patients). We conducted a paired t-test to evaluate change in knowledge scores and used generalized estimating equation-based (GEE) models with link function of Poisson distribution and an exchangeable correlation structure to compare referral outcomes. The models included exposure to training (Yes/No), pre- and post-training time periods and the interaction of these two indicators as predictors. All analyses were two-sided, statistical significance was set at type I error of 5% and analyses were conducted using R Statistical Software.